CLINICAL TRIAL: NCT03547960
Title: The Use of Soluble Fibre for the Prevention of Gestational Diabetes Among High-risk Women. A Pilot Study.
Brief Title: Effect of Fibre Supplements on Gestational Diabetes
Acronym: GG-GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRAS ID: 230813
Record Dates: First submitted 2018-05-10; First posted 2018-06-06 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — guar gum; Cellulose

STUDY DESIGN:
Intervention Model Description: Open label controlled study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guar gum (intervention) (Experimental): 5 g of Guar gum fibre supplement with meals three times a day (total daily 15 g) for 12 weeks
  Interventions: Dietary Supplement: Guar gum
- Control/Cellulose (Placebo Comparator): 5 g of Cellulose fibre supplement with meals three times a day (total daily 15 g) for 12 weeks
  Interventions: Dietary Supplement: Cellulose

INTERVENTIONS:
Dietary Supplement: Guar gum — Fibre supplement to be taken with each meal
  Arms: Guar gum (intervention)
Dietary Supplement: Cellulose — Placebo. Fibre supplement to be taken with each meal
  Arms: Control/Cellulose

SUMMARY:
The primary aim of this study is to evaluate the effect of a soluble fibre supplement in the development of gestational diabetes in women at high-risk. The secondary aim will be to evaluate the effect of the soluble fibre supplement on glycaemic control in high-risk women who develop gestational diabetes in early pregnancy.

DESIGN The study plans to conduct a randomised open label controlled study to evaluate the effect of the consumption of soluble fibre, from early to mid-pregnancy, on the incidence of gestational diabetes, insulin sensitivity, insulin secretion and metabolic control in GDM diagnosed participants.

POPULATION The study team will be studying women with diagnosis of gestational diabetes in previous pregnancies, (considered as high-risk) aged >18 years.

TREATMENT Participants in the treatment arms will be 5 gr of Guar gum fibre supplement with meals three times a day (total daily 15 g). Participants in the placebo arms will be taking 5 gr of Cellulose three times a day (total daily dose 15 g).

DURATION Participants will be involved for 12 weeks.

OUTCOMES Primary outcome: In women with 16-week negative OGTT, GDM at 28 weeks

DETAILED DESCRIPTION:
Aim: To evaluate the effect of a soluble fibre supplement in glucose metabolism in pregnant women at high risk of developing gestational diabetes.

Study methodology: 12 week randomised, placebo-controlled, single-blinded study.

Intervention: Women will first be categorised according to their glycaemic status into two groups: GDM and glucose tolerant women. Afterwards, each group will be randomised into two groups and given either

1. Fibre supplement (Guar gum)
2. Placebo (Cellulose) The participants will take the dietary supplement three times a day for 12 weeks. They will receive regular antenatal control according to NICE guidelines recommendations. Compliance will be addressed by weekly phone calls.

   Number of volunteers: The number of participants will be arbitrarily define as no data of this type of intervention exists in this cohort. 60 participants will be recruited. Previous studies, outside pregnancy, have observed metabolic effects in samples of 15-40 subjects.

   Recruitment: Women will be recruited in the antenatal clinic at Queen Charlotte and Chelsea's Hospital. An information sheet will be provided to eligible women in the first antenatal visit to explain the purposes of the study. Women who decide to take part will be asked to sign a consent form.

   Randomisation: Initially women will be categorised according to glycaemic status in two cohorts: Glucose tolerant and Early gestational diabetes (GDM) cohort. Each of the two cohorts will then be independently randomised to either intervention or standard care using the sealed envelope website. Guar gum (intervention) and cellulose (placebo) will be provided in identical packed sachets.

   PRIMARY OUTCOME MEASURES
   * GDM at 28 weeks
   * Glucose values at 0 and 120 minutes during an OGTT performed at 28 weeks in the glucose tolerant group.

   SECONDARY OUTCOME MEASURES

   Assessing insulin sensitivity and insulin secretion at 28 weeks of pregnancy in the glucose tolerant cohort of women through validated indices using glucose and insulin (or C-peptide) values derived from the OGTT.
   * Insulin sensitivity will be assessed using the Matsuda formula
   * Insulin secretion will be assessed by second-void fasting UCPCR.

     6. ASSESSMENT AND FOLLOW UP Women will be assessed by the researchers at four different visits. At the first antenatal visit, the general care team will mentioned the study, if the patient consents, she will then be approached by the researchers to explain the study protocol. At the second visit, when the OGTT is performed, women who decided to take part in the study will sign the consent from. At the next antenatal visit where results from the OGTT are explained, women included will be randomised. The last research visit will take place at 28 weeks gestation. Additionally, they will be contacted weekly, by telephone to assess compliance and confirm willingness to participate in the study.
     1. st visit (≤16 weeks gestation) Women with a previous history of GDM will be considered at high risk of recurrence and will be referred to the antenatal clinic before 16 weeks of pregnancy. At this first visit, an information sheet will be provided and women will have time to consider if they are willing to participate and inform the research team at their next antenatal visit.
     2. nd visit Women who decide to participate will inform the research team when they attend their second antenatal visit, when an OGTT is to be performed. I After the participants have agreed to take part in the study and consent has been signed, data regarding anthropometrics, demographics and medical history will be collected. This information will be obtained by reviewing the participant's medical notes.
     3. rd visit (Randomisation)

        After obtaining the results from the OGTT, women will be categorised by their glycaemic status and divided into two independent cohorts:
   * Women diagnosed with gestational diabetes (according to NICE guidelines 2015 diagnostic criteria): early GDM cohort
   * Women with normal glucose tolerance or impaired glucose tolerance but not fulfilling GDM criteria: Glucose tolerant cohort.

   Women from each cohort will be randomised into two groups after the results of the OGTT are obtained:
   * Intervention group: Guar gum fibre supplement
   * Placebo group: Cellulose supplement Women will the fibre supplement 3 times a day (with each main meal) until the 28th week of pregnancy when they will be re-evaluated.

     4rd visit (28th weeks gestation)

   Glycaemic status will be assessed at 28 weeks gestation in the two cohorts of women participating in the study:
   * Women from the Glucose tolerant cohort will undergo a second OGTT.
   * In women in the Early GDM cohort, glycaemic control will be assessed by the need of insulin treatment (yes/no).

   PROCEDURES Women will be advised to fast for 10 hours the night before the oral glucose tolerance test. They will also be advised no to restrict carbohydrate ingestion the three days prior to the OGTT. At the antenatal clinic, blood samples will be collected at baseline (0 min) and at 120 min after the administration of an oral load of 75 g of glucose.

   Serum insulin and C-peptide will be collected at 0 and 120 min during the OGTT.

   ASSESSMENTS

   (i) Gestational diabetes Gestational diabetes will be diagnosed if fasting plasma glucose >5.6 mmol/L and/or 120 min plasma glucose >7.8 mmol/L after the glucose load administered in the OGTT. Women with fasting plasma glucose <5.6 mmol/L and 120 min plasma glucose <7.8 mmol/L will be classified as "Glucose tolerant".

   (ii) Insulin sensitivity Insulin sensitivity will be assessed using the Matsuda index as originally described (18) (Equation 1) and using two modified Matsuda equations in which insulin is substitute by either serum or urinary C-peptide (21,22) (Equations 2 and 3).

   Equation 1. ISOGTT= 10,000 / √ {[FPG x fasting insulin] x [mean glucose x mean insulin during OGTT]} Equation 2. ISOGTTC-pep=500,000/√{[FPGxFsC-pep] x [mean glucose x mean sC-pep during the OGTT]} Equation 3. ISOGTT-UCPCR=500,000/√{[FPG×FUCPCR pmol/mmol] x [mean glucose x mean UCPCR during the OGTT]}

   (iii) Insulin secretion Insulin secretion will be estimated by the UCPCR obtained using the fasting second-void urine sample, as it is strongly correlated with serum insulin, serum C-peptide (19) and 24-h urinary C-peptide (20).

   Insulin response will be estimated using the UCPCR calculated with 120 min post-OGTT urine sample, as it is strongly correlated with the C-peptide and insulin area under the curve (19).

   (iv) Need of insulin treatment, Days to insulin treatment and Total insulin dose Medical records of women in the Early GDM cohort will be review in order to determine the need of insulin treatment (yes/no) at 28 weeks gestation.

   WITHDRAWAL CRITERIA Participants will be free to withdraw at any time and are not required to give a reason.

   STATISTICS AND DATA ANALYSIS Data handling and analysis will be carried out by SPSS version 20.0 version. No power calculation to decide sample size will be used. The number of participants has been arbitrarily defined, as it is a pilot study. The study aims to recruit 40 women.

   In the Glucose tolerant women cohort:

   For the primary outcome, GDM (yes/no), logistic regression analysis will be performed.

   For the secondary outcomes, insulin sensitivity and insulin secretion, linear regression analysis will be performed.

   In the early GDM cohort:

   For the primary outcome, need for insulin treatment (yes/no), logistic regression analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of GDM in previous pregnancies
* Age ≥ 18 years
* Singleton pregnancy
* ≤ 16 weeks gestation

Exclusion Criteria:• Women unable or unwilling to give consent

* Pre-gestational diabetes or use of anti-diabetic medication in the first visit
* Significant chronic medical conditions (cardiovascular, liver or kidney disease)
* Women participating in other medical trial
* Women who have undergone bariatric surgery
* Women with milk allergy/intolerance
* Women unable to speak/understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 60 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, PhD, Principal Investigator — Chair of Nutrition. Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Guar Gum: 5 g of Guar gum fibre supplement with meals three times a day (total daily 15 g) for 12 weeks
  Guar gum: Fibre supplement to be taken with each meal
Period: Overall Study
Arm/Group | Guar Gum | Control/Cellulose
Started | 30 | 30
Completed | 10 | 10
Not Completed | 20 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guar Gum | Control/Cellulose | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (4.8) | 32.6 (4.4) | 34.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5 | 6 | 11
  Non-caucasian | 17 | 13 | 30
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Numbers Diagnosed With Gestational Diabetes
Description: An Oral glucose tolerance test will be performed. Gestational diabetes will be diagnosed if fasting plasma glucose >=5.3 and or 120 min plasma glucose >=7.8
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Guar Gum | Control/Cellulose
Number analyzed (Participants) | 10 | 10
Participants | 7 | 6
Statistical Analysis 1: Comparison: Guar Gum; Test type: Superiority; p = 0.639, Chi-squared
Statistical Analysis 2: Comparison: Guar Gum; Test type: Superiority; p = 0.283, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Comparison of Insulin Sensitivity Between the 2 Experimental Groups (Gur and Cellulose Groups)
Description: Insulin sensitivity will be assessed using the Matsuda index (is an whole body insulin sensitivity index that reflects a composite estimate of hepatic and muscle insulin sensitivity) in line with the following modified Matsuda equation in which insulin is substituted by the serum concentration of C-peptide for estimation purposes. In the the above index scale a lower number indicates lower sensitivity.
  Equation: ISOGTTC-pep=500,000/√{[FPGxFsC-pep] x [mean glucose x mean sC-pep during the OGTT]} There is no maximum or minum
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guar Gum | Control/Cellulose
Number analyzed (Participants) | 22 | 19
score on a scale | 269.7 (141.6) | 324.2 (210.3)

3. Secondary Outcome: Comparison of Insulin Secretion Between the 2 Experimental Groups (Guar and Cellulose)
Description: HOMA-IR is a model that uses the static concentrations of fasting glucose and insulin for determination of insulin resistance and pancreatic beta-cell function. In the the above model scale a lower number indicates lower secretion.
  The validity of HOMA-IR index is lower in patients with low body mass index (BMI), low-activity of beta cells and high levels of blood glucose Homa IR =fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5. There is no maximum or minimum
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Guar Gum | Control/Cellulose
Number analyzed (Participants) | 22 | 19
score on a scale | 433.9 (377.5) | 479.8 (508.8)
Statistical Analysis 1: Comparison: Guar Gum; Test type: Superiority; p = 0.564, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Guar Gum | Control/Cellulose
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 11/22 | 8/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guar Gum (N=22) | Control/Cellulose (N=19)
Abdominal discomfort (Gastrointestinal disorders) | 11 (11) | 8 (8) — Abdominal discomfort, flatulence, abdominal distension

LIMITATIONS AND CAVEATS:
Recruitment was difficult during the COVID period We have a high dropout rate. Women diagnosed with early GDM abandoned the study after diagnosis and withdrew consent so their data is not analysed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT03547960/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03547960/ICF_001.pdf